CLINICAL TRIAL: NCT04504071
Title: Dacomitinib in Advanced Non-small Cell Lung Cancer Patients With Uncommon EGFR Mutations: A Single Center and Exploratory Study
Brief Title: Dacomitinib in Lung Cancer With Uncommon EGFR Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, director of respiratory department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS2034
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer Metastatic; EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dacomitinib Arm (Other): This is a single arm study.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Patients will receive continuous oral therapy with the study drugs (dacomitinib 45 mg) until disease progression or unacceptable toxicity.

SUMMARY:
This is a single center and exploratory study, aiming to analyze the efficacy and safety of dacomitinib-a pan-HER and irreversible TKI in subjects with diagnosed stage IIIB/IV or recurrent NSCLC. All subjects will have tumors that test positive for at least one uncommon EGFR activating mutation (do not have drug-resistant pattern, e.g. 20 insertion or 20T790M). All patients will be of histo- and/or cytopathology confirmed. Determination of the EGFR mutation type will be performed in the pathological department of Shanghai Chest Hospital. Both ARMS method or targeted sequencing are acceptable. It is not acceptable for subjects with the presence of the exon 20T790M mutation or insertion together with either EGFR activating mutations (exon 19 deletion or the L858R mutation in exon 21) or uncommon EGFR mutations. 10ml peripheral blood must be available for concomitant study. All eligible subjects must have adequate renal, hepatic, and hematologic function, as defined in "inclusion criteria".

Patients will receive continuous oral therapy with the study drugs (dacomitinib 45 mg) until progressive disease as defined by RECIST version 1.1 or judged by investigator that the patient no longer derives clinical benefit from study treatment. At the time of progression and removal from study treatment, the subject may receive any regulatory approved therapy at the judgment of the investigator. Timely and complete disease assessments in this study are important. Every effort should be made to ensure disease assessments performed as scheduled to prevent the introduction of bias into the assessment of efficacy. Failure to perform any of the required disease assessments will result in the inability to determine disease status for that time point. Frequent off schedule or incomplete disease assessments have the potential to weaken the study conclusion.

Subjects who have progressive disease per RECIST version 1.1 confirmed by the investigator believes it is in their best interest to continue on their study therapy, will be allowed to continue on their therapy with or without local therapy (e.g. surgical removal and/or radiation of a single lesion), at the discretion of the investigator until any alternate or additional systemic anti-cancer therapy regimen is implemented. The subsequent new cancer therapy (including, for systemic therapy, drugs administered, date of initiation and discontinuation of each drug) and OS will be recorded. Each subject will be followed for survival status and subsequent cancer therapies up to 48 months from the date of first dosing. This data may be collected from subjects by telephone, and if collected should be entered into the CRF.

ELIGIBILITY:
Inclusion criteria: Only patients who meet all of the following criteria will be enrolled into this study:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with locally advanced (stage III B/III C), metastatic or recurrent (stage IV) NSCLC confirmed by histology or cytology who are unable to undergo surgery and radical concomitant radiochemotherapy and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. Patients harboring uncommon EGFR mutations. Uncommon EGFR mutations were defined as mutations in exon 18-21 but except for 19del, 21L858R and well-established drug resistant type (20 insertion, 20T790M, 19L747S, 19L747P, D761Y, 21T854A). Mutations should be previously reported that it was sensitive to first- or second-generation TKIs. Detailed mutation type including:

   Mutation in exon 18:

   G719X(X=A/C/S/D/E), 18del, E709X(X=G/M/V/H/DA/K), V689M, S720P/F, P699S, N700D, E709Q, G721A, V740A, L718P;

   Mutation in exon 19:

   Few exon 19 point mutations with unknown structure and kinase activity have been found in EGFR-TKI responders, however, a new class of sensitizing mutations, exon 19 insertions, were recently found, these patients were also eligible for this study: I744_K745insKIPVAI, K745_E746insIPVAIK, K745_E746insVPVAIK, K745_E746insTPVAIK.

   Mutation in exon 20:

   Including S768I, V765A, T783A, V774A, S784P, R776C, R776H, V765M, G779C, G779F, G779S, T783A, T783I, L798F, L798H, K806E, Q812R, L814P

   Mutation in exon 21:

   L861Q, R831H, V834I, L838P, L861R.

   Others:

   Patients with complex mutation but do not have drug-resistant pattern (e.g. 18G719A+20S768I, 18 E709X+21L861Q) are also eligible. However, individuals who have common mutation (e.g. 19del+21L861Q, 18G719X+21L858R) were not eligible.
3. Age ≥18 years and ≤75 years;
4. ECOG PS score: 0 to 2
5. Previously untreated with EGFR-TKIs including first-, second- or third generation agents. Subjects who were only treated with chemotherapy were eligible. Patients who have received adjuvant chemotherapy but disease recurrence must have happened at least 6 months after the last dose of chemotherapy. Palliative radiotherapy must be completed 7 days before the first dose of study drugs;
6. The main organs function is normal, that is, the following criteria met:

   * Good hematopoietic function, defined as absolute neutrophil count ≥1.5×109 /L, platelet count≥100 ×109 /L, hemoglobin ≥90g/L [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment]
   * Biochemical test results should meet the following criteria: BIL < 1.25 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Cr ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; Coagulation function is good, INR and PT ≤1.5 times ULN; if the subject is receiving anticoagulant treatment, PT should be within the prescribed range of use of anticoagulant drugs;
7. Women of child-bearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; non-breast-feeding patients whose serum or urinary pregnancy test should be negative; male patients should agree to take contraceptive measures during the study and within 6 months after the study.
8. Patients are voluntarily enrolled into the study, sign the informed consent form and have good compliance.

Exclusion criteria

Patients who meet any of the following criteria will be excluded:

1. Small cell lung cancer (including mixed small cell and non-small cell lung cancer);
2. Patients who have received EGFR-TKIs as adjuvant or salvaged treatment;
3. Patients with 19del or 21L858R or well-established drug resistant type (20 insertion, 20T790M, L747S, L747P, D761Y, T854A).
4. Patients with many factors affecting oral medication, such as dysphagia, gastrointestinal resection, chronic diarrhea and intestinal obstruction;
5. Patients who are known to have brain metastases including asymptomatic metastasis, spinal cord compression, carcinomatous meningitis, or brain or leptomeningeal disease diagnosed by CT or MRI at the time of screening;
6. Patients with severe and / or uncontrolled diseases, such as:

   * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; uncontrolled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
   * Active or uncontrolled serious infection;
   * Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
   * Not completely controlled eye inflammation or eye infection, or any condition that may lead to the above-mentioned ocular diseases
   * Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
   * Routine urine test result indicates that urine protein ≥++, and 24-hour urine protein quantitation is confirmed to be > 1.0 g;
   * Active tuberculosis, etc.;
   * Uncontrolled hypercalcemia (> 1.5 mmol/L calcium ion or calcium > 12 mg/dL or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued diphosphate therapy;
   * Long-term unhealed wounds or fractures;
7. Patients who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders;
8. Patients who are known to have severe allergies (≥ grade 3) to active ingredients and any excipients of dacomitinib
9. Patients who have other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) at the same time; patients who are evaluated by the investigator to have concomitant diseases that seriously endanger the safety of the patients or affect the patients completing the study.
10. The subjects or their sexual partners cannot or refuse to take effective contraceptive measures during the clinical trial
11. Pregnant or breast-feeding women
12. Patients in other situations who are evaluated by the investigator to be ineligible to be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate （ORR） | 6-12 weeks
  ORR was defined as the proportion of patients with a complete response (CR) or partial response (PR) per the investigator's assessment using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Disease control rate | 6-12 weeks
  The disease control rate (DCR) was defined as the sum of the proportions of patients who had CR, PR, and stable disease (SD) using RECIST 1.1 criteria
PFS | 13-15months
  PFS was defined as the time from study treatment initiation to the first occurrence of documented disease progression or death from any cause during the study, whichever occurred first.
Overall survival | 22-25months
  OS was defined as the time from the first dose of study treatment to the time of death from any cause during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang B, Shi C, Gao Z, Zhong H, Xiong L, Gu A, Wang W, Chu T, Zhang W, Wang H, Zhang X, Zhong R, Han B. Rationale and design of a phase II trial of dacomitinib in advanced non-small cell lung cancer patients with uncommon epidermal growth factor receptor mutations: a prospective and single arm study (DANCE study). BMC Cancer. 2022 Mar 19;22(1):294. doi: 10.1186/s12885-022-09409-3. PMID 35305596